CLINICAL TRIAL: NCT02112643
Title: Selenium - ITEDS: A North American Study
Brief Title: Selenium in Mild Thyroid Eye Disease in North America
Acronym: S-ITEDS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Collaborators: International Thyroid Eye Disease Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAL9502
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Associated Ophthalmopathies
Keywords: Thyroid eye disease; Thyroid orbitopathy; Graves' orbitopathy; Graves' ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Selenic Acid; Selenium; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selenium (Active Comparator): 100 micrograms of sodium selenate will be taken orally twice daily (total 200 micrograms daily) for 6 months.
  Interventions: Drug: Sodium selenate
- Sugar pill (Placebo Comparator): A placebo pill will be taken orally twice daily for 6 months.
  Interventions: Dietary Supplement: Sugar pill

INTERVENTIONS:
Drug: Sodium selenate — A 100 microgram pill will be orally administered twice a day for 6 months.
  Other Names: Selenium
  Arms: Selenium
Dietary Supplement: Sugar pill — The placebo pill will be constructed to look exactly like the selenium pill, but will have no active ingredients. This will be orally administered for 6 months.
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether sodium selenite is helpful in the treatment of mild thyroid eye disease in North America.

DETAILED DESCRIPTION:
Thyroid eye disease (TED) is a disease in which the soft tissues surrounding the eye can become inflamed, scarred, and at times permanently damaged in an autoimmune reaction highly associated with abnormal thyroid hormone levels. Some patients have much more severe TED than others, but overall, most patients reach a point with relatively stable TED after 1 to 2 years. A recent European study showed that oral selenium, a trace mineral involved in anti-oxidation and immune regulation, could actually alter the course of mild TED, lessening its signs and symptoms and even improving the quality of life of those who took it. The investigators would like to perform a sister study throughout North America. In this randomized, double-blinded, multi-center trial, some subjects with mild TED would be given 100 micrograms of sodium selenite twice a day; others would receive a placebo. Signs, symptoms, and quality of life would be measured at regular intervals throughout the 6 month period of drug administration, and for 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide informed consent
* Able to swallow pills
* Mild thyroid eye disease requiring no past treatment other than ophthalmic drops or ointment
* Euthyroid: at least 2 months if on medication irregardless of thyroidectomy status; at least 6 months after radioiodine therapy; if euthyroid for the year prior to enrollment, needs normal thyroid-stimulating hormone (TSH) within last 3 months; if uncontrolled for the year prior to enrollment, needs normal TSH and free T4 within last 3 months; if TSH low, needs normal T3 and free T4
* If you are currently taking any selenium supplementation, you will be asked to discontinue its usage, "wash out", for 1 month before you are enrolled.

Exclusion Criteria:

* Moderate or severe thyroid eye disease (based upon International Thyroid Eye Disease Society VISA form), including: grade 2 chemosis or lid edema; corneal exposure with threat of or resulting in perforation; optic neuropathy; grade 3 restriction of any extraocular muscle
* Double vision (diplopia) in primary or reading positions
* Duration of thyroid eye disease greater than 12 months (as per patient history)
* Drug or alcohol abuse
* Severe systemic illness (defined by treating physician)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Estimated); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Difference in Quality of Life score | Six months
  Using GO-QOL score
Difference in Quality of Life score | Twelve months
  GO-QOL score
Change in Thyroid Eye Disease | Six months
Change in Thyroid Eye Disease | Twelve months

SECONDARY OUTCOMES:
Difference in Clinical Activity Score | Six months
Difference in Clinical Activity Score | Twelve months
Difference in Quality of Life score | Six months
  TED-PRO
Difference in Quality of Life score | Twelve months
  TED-PRO
Difference in Quality of Life score | Six months
  TED-QOL
Difference in Quality of Life score | Twelve months
  TED-QOL
Difference in development of optic neuropathy | Twelve months
Difference in Inflammatory Index | Six months
  Improvement
Difference in Inflammatory Index | Twelve months
  Improvement
Difference in Inflammatory Index | Six months
  Deterioration
Difference in Inflammatory Index | Twelve months
  Deterioration
Difference in diplopia score | Six months
  Improvement
Difference in diplopia score | Twelve months
  Improvement
Difference in diplopia score | Six months
  Deterioration
Difference in diplopia score | Twelve months
  Deterioration
Difference in degrees of restriction | Six months
  Improvement
Difference in degrees of restriction | Twelve months
  Improvement
Difference in degrees of restriction | Six months
  Deterioration
Difference in degrees of restriction | Twelve months
  Deterioration
Difference in exophthalmos scores | Six months
  Improvement
Difference in exophthalmos scores | Twelve months
  Improvement
Difference in exophthalmos scores | Six months
  Deterioration
Difference in exophthalmos scores | Twelve months
  Deterioration
Difference in eyelid aperture | Six months
  Improvement
Difference in eyelid aperture | Twelve months
  Improvement
Difference in eyelid aperture | Six months
  Deterioration
Difference in eyelid aperture | Twelve months
  Deterioration

OTHER OUTCOMES:
Fasting glucose level | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Kazim, MD, Principal Investigator — International Thyroid Eye Disease Society

REFERENCES:
- [Background] Marcocci C, Kahaly GJ, Krassas GE, Bartalena L, Prummel M, Stahl M, Altea MA, Nardi M, Pitz S, Boboridis K, Sivelli P, von Arx G, Mourits MP, Baldeschi L, Bencivelli W, Wiersinga W; European Group on Graves' Orbitopathy. Selenium and the course of mild Graves' orbitopathy. N Engl J Med. 2011 May 19;364(20):1920-31. doi: 10.1056/NEJMoa1012985. PMID 21591944
- See also: This is the International Thyroid Eye Disease Society (ITEDS) website. — http://thyroideyedisease.org/